CLINICAL TRIAL: NCT01021358
Title: A Phase 1 Study to Assess the Effect of Ketoconazole on the Pharmacokinetics of ABT-263 (Navitoclax)
Brief Title: A Study to Assess the Effect of Ketoconazole on the Metabolism of ABT-263 (Navitoclax).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Andrew Krivoshiik, MD, PhD, Medical Director, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-957
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-12

CONDITIONS: Lymphoma; Chronic Lymphocytic Leukemia; Solid Tumors
MeSH Terms: conditions — Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — navitoclax; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (ABT-263 and Ketoconozole) (Experimental)
  Interventions: Drug: ABT-263; Drug: Ketoconazole

INTERVENTIONS:
Drug: ABT-263 — Subjects will be dosed with ABT-263, then dosed with ABT-263 in combination with Ketoconazole.
Drug: Ketoconazole — Subjects will be dosed with ABT-263, then dosed with ABT-263 in combination with Ketoconazole.

SUMMARY:
This is a single dose, open-label, single or multiple center study to determine the interaction of ketoconazole with ABT-263 in approximately 12 subjects with cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Has a non-hematologic malignancy (radiographic, histologic, or cytologic confirmation), or hematologic malignancy (histologic or cytologic confirmation) that is either: relapsed or refractory to standard therapy, failed at least one prior therapy or no known effective therapy exists.
* In the investigator's opinion, the subject's life expectancy is at least 90 days.
* If clinically indicated, (e.g., subjects over the age of 70) subjects must have documented brain imaging (MRI or CT) negative for subdural or epidural hematoma within 28 days prior to the first dose of study drug.
* Subjects with brain metastases must have clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function and no evidence of CNS disease progression as determined by CT or MRI within 21 days prior to the first dose of study drug.

Exclusion Criteria:

* History of or is clinically suspicious for cancer-related central nervous system (CNS) disease.
* Has undergone an allogeneic stem cell transplant.
* Has an underlying, predisposing condition of bleeding or currently exhibits signs of bleeding.
* Has active peptic ulcer disease or other hemorrhagic esophagitis/gastritis.
* Has active immune thrombocytopenic purpura or a history of being refractory to platelet transfusions (within 1 year prior to the first dose of study drug).
* Significant history of cardiovascular disease (e.g., MI, thrombotic or thromboembolic event in the last 6 months), renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease. Female subject is pregnant or breast-feeding.
* History of or an active medical condition(s) that affects absorption or motility (e.g., Crohn's disease, celiac disease, gastroparesis, short bowel syndrome, etc).
* Exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to: active systemic fungal infection; diagnosis of fever and neutropenia within one week prior to study drug administration.
* Received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal (with the exception of hormones for hypothyroidism or estrogen replacement therapy [ERT], or agonists required to suppress serum testosterone levels [e.g., LHRH, GnRH, etc.] for subjects with prostate cancer
* Currently receiving or requires anticoagulation therapy or any drugs or herbal supplements that affect platelet function.
* Currently receiving or requires anti-fungal treatment or CYP3A inhibitors. In the opinion of the Investigator, the subject is an unsuitable candidate to receive ABT-263.
* History of or is clinically suspicious for cancer-related central nervous system (CNS) disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To determine the effect of ketoconazole on the pharmacokinetics of ABT- 263. | Weekly

SECONDARY OUTCOMES:
To determine the safety of ABT-263 when administered alone and in combination with Ketoconazole in these patients. | Daily

CONTACTS AND LOCATIONS:
Locations (1):
- Site Reference ID/Investigator# 25068, San Antonio, Texas, United States